CLINICAL TRIAL: NCT00530088
Title: Photodynamic Therapy With Photofrin® for Treatment of Dysplasia, Carcinoma In Situ and Stage I Carcinoma of the Oral Cavity and the Larynx: A Pilot Study
Brief Title: Photodynamic Therapy Using Porfimer Sodium in Treating Patients With Recurrent Mouth or Throat Dysplasia or Recurrent In Situ Cancer or Stage I Cancer of the Mouth or Throat
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: new competing studies
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000564841; RPCI-RPC-01-08 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-06

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage 0 laryngeal cancer; stage 0 lip and oral cavity cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Laryngeal Neoplasms; Mouth Neoplasms | interventions — Dihematoporphyrin Ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Porfimer Sodium (Experimental): Patients receive porfimer sodium subcutaneously followed by photodynamic therapy (PDT) comprising laser light delivered by a single or a diffuser (i.e., for broad areas of dysplasia) fiberoptic lens fiber.
  Interventions: Drug: porfimer sodium; Drug: Photdynamic Therapy (PDT)

INTERVENTIONS:
Drug: porfimer sodium — IV
Drug: Photdynamic Therapy (PDT)

SUMMARY:
RATIONALE: Photodynamic therapy uses a drug that becomes active when it is exposed to a certain kind of light. When the drug is active, tumor cells are killed. Photodynamic therapy using porfimer sodium may be effective against mouth or throat dysplasia and cancer of the mouth and throat.

PURPOSE: This phase I trial is studying how well photodynamic therapy using porfimer sodium works in treating patients with recurrent mouth or throat dysplasia, recurrent in situ cancer of the mouth or throat, or stage I cancer of the mouth or throat.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the response of patients with recurrent dysplasia, squamous cell carcinoma in situ, or stage I squamous cell carcinoma of the oral cavity or the larynx treated with photodynamic therapy using porfimer sodium.
* To identify the local toxicity of this treatment in these patients.

OUTLINE: Patients receive porfimer sodium subcutaneously followed by photodynamic therapy (PDT) comprising laser light delivered by a single or a diffuser (i.e., for broad areas of dysplasia) fiberoptic lens fiber. Patients with incompletely treated or missed sites of disease may receive another dose of laser light on day 5 without additional porfimer sodium. Patients with multicentric disease may undergo additional PDT at least 4-6 weeks after the initial treatment.

After completion of study therapy, patients are followed for 1-2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy confirmed oral cavity or larynx lesion with mild-to-severe dysplasia OR in situ or stage I (T1, N0) squamous cell carcinoma of the oral cavity or larynx
* Recurrent disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* WBC ≥ 4,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 2.0 mg/dL
* Creatinine ≤ 2.0 mg/dL
* Alkaline phosphatase ≤ 3 times upper limit of normal (ULN)
* SGOT ≤ 3 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must practice effective contraception
* No porphyria or hypersensitivity to porphyrin or porphyrin-like compounds

PRIOR CONCURRENT THERAPY:

* Any type of prior therapy allowed
* More than 4 weeks since prior and no concurrent chemotherapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2001-10; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nestor R. Rigual, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Result] Rigual NR, Thankappan K, Cooper M, Sullivan MA, Dougherty T, Popat SR, Loree TR, Biel MA, Henderson B. Photodynamic therapy for head and neck dysplasia and cancer. Arch Otolaryngol Head Neck Surg. 2009 Aug;135(8):784-8. doi: 10.1001/archoto.2009.98. PMID 19687399

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Porfimer Sodium
Started | 30
Completed | 20
Not Completed | 10
Not completed — Disease Progression | 4
Not completed — Physician Decision | 4
Not completed — Other Not Specified | 2

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Porfimer Sodium
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Response Rate 9.0 TUMOR RESPONSE 9.1 Tumor response will be evaluated at each follow-up visit. 9.2 Objective Tumor Response 9.21 Complete Response - CR1 Complete absence of visible lesion and negative biopsy. CR2 Complete absence of visible lesions without biopsy. 9.22 Partial Response. Reduction in the lesion size by 50% or more in the maximum size of the initial lesion or reduction in grade of lesion, e.g. severe -> mild dysplasia. Patients that have any physical evidence of residual leukoplakia or erythroplasia will require biopsy.
  9.23 No Response. All responses less than a Partial Response are considered as No Response.
  9.24 Progressive Disease. Any increase in size of the treated lesion or an increase in grade of the treated lesion, i.e. mild to severe dysplasia.
Time Frame: 2 years
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Porfimer Sodium
Number analyzed (Participants) | 29
percentage of participants | 3.5 [0 to 10]

2. Primary Outcome: Local Toxicity
Description: Number of patients with an adverse event
Time Frame: 30 days
Population: All treated and eligible patients
Measure: Number; unit: participants
Arm/Group | Porfimer Sodium
Number analyzed (Participants) | 30
participants | 29

ADVERSE EVENTS:
Arm/Group | Porfimer Sodium
Serious Adverse Events (participants affected / at risk) | 3/30
Other Adverse Events (participants affected / at risk) | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Porfimer Sodium (N=30)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Porfimer Sodium (N=30)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Lip oedema (Gastrointestinal disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 2 (2)
Oedema mouth (Gastrointestinal disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 4 (5)
Oral pruritus (Gastrointestinal disorders) | 1 (1)
Face oedema (General disorders) | 2 (2)
Oedema (General disorders) | 14 (15)
Pain (General disorders) | 16 (18)
Herpes virus infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 18 (21)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the study's early termination, as a result of new competing studies, target accrual was not reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes